

| IRAS ID: |
|----------|
|----------|

Study Number:

Participant Identification Number for this trial:

## **CONSENT FORM**

Title of Project: Surgical Techniques: Robotic versus conventional Laparoscopic cholecystectomy IN benign Gallbladder disease.

| Name | e of Researcher: | | | |
|---|---|---|---|---|
| | | | Ple | ase initial box |
| 1. | I confirm that I have read the information sheet dated (version.1.1) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | | | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | | | |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | | | |
| 5. | I agree to my General Practitioner being informed of my participation in the study. | | | |
| 6. | I understand that the information held and maintained by Portsmouth Hospitals Univerity NHS Trust may be used to help contact me or provide information about my health status. | | | |
| 7. | I agree to take part i | n the above study. | | |
| Name of Participant | | Date | Signature | |
| Name of Person seeking consent | | Date | Signature | |